CLINICAL TRIAL: NCT03607253
Title: Investigating the Gender-related Response of Muscle Fatigue of the Medial Longitudinal Arch Height in Healthy Young
Brief Title: Muscle Fatigue and Foot Biomechanics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Trakya University (Other)
Responsible Party: Principal Investigator, Halit SELÇUK, Principal Investigator, Trakya University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: TUTF-BAEK 2018/159
Record Dates: First submitted 2018-07-19; First posted 2018-07-31 (Actual); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Foot, Flat
Keywords: medial longitudinal arch; foot
MeSH Terms: conditions — Flatfoot

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Men (Other): Healthy young men aged between 18-25 years
  Interventions: Other: repetitive heel rise activity
- Women (Other): Healthy young women aged between 18-25 years
  Interventions: Other: repetitive heel rise activity

INTERVENTIONS:
Other: repetitive heel rise activity — Participants will perform a maximal number of single-legged heel rises on a 10 degrees incline board. Participants will be permitted to apply for fingertip support at shoulder height on a wall in front of them. The test will be terminated when participants could no longer lift their heels from the incline board. The number of correct heel rises will be counted for each leg and will be used as Heel Rise Test score.

SUMMARY:
Medial longitudinal arch (MLA) is a curve of the foot located at the medial side of the body and protection of the height of the MLA is an important factor for limb health.

This study was planned with the aim of investigating the response of the MLA height to the repetitive muscle activity and determine the gender-related differences.

ELIGIBILITY:
Inclusion Criteria:

* healthy young females and males who want to participate to the study

Exclusion Criteria:

* have orthopedic, physiologic, psychiatric, neurologic or systemic disorders
* have present medication

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — females and males
Enrollment: 60 (Actual)
Dates: Start 2018-09-30 (Actual); Primary Completion 2018-10-15 (Actual); Study Completion 2018-10-30 (Actual)

PRIMARY OUTCOMES:
Navicular Drop | at first minute, change from baseline arch height at 2nd minutes
  Vertical distance of navicular tuberosity (highest point of the MLA) to the ground is measured for two times. First; with the foot placed in subtalar joint neutral position in full weight-bearing and second; in relaxed standing position. The difference between the two values are recorded as Navicular Drop (mm).

CONTACTS AND LOCATIONS:
Locations (1):
- Trakya University, Edirne, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided